CLINICAL TRIAL: NCT01443585
Title: Clinical Performance Evaluation of a Progressive Addition Lens Among Presbyopic Patients
Brief Title: Clinical Evaluation of a Progressive Addition Lens (PAL)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PALsCTIL
Record Dates: First submitted 2011-09-14; First posted 2011-09-29 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2011-09

CONDITIONS: Presbyopia
Keywords: Progressive Addition Lens; Multifocal; Presbyopia
MeSH Terms: conditions — Presbyopia | interventions — Eyeglasses

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Progressive Addition Lens (Shamir PrimeIITM) Spectacles — A pair of progressive addition lenses manufactured according to the subject's personal prescription.

SUMMARY:
The purpose of the trial is to clinically evaluate the performance of a progressive addition lens among presbyopic patients.

This evaluation will be done by performing visual tests and collecting subjective information from subjects wearing the lens which will be manufactured according to personal prescription.

ELIGIBILITY:
Inclusion Criteria:

* An ability to comprehend and give an informed consent for participation in the trial
* Presbyopia

Exclusion Criteria:

* Concurrent participation in another clinical trial
* Age<18
* For female subjects: pregnancy \ planning a pregnancy \ lactating at the time of enrollment
* Imbalanced diabetes \ high blood pressure \ thyroid disease
* Infectious disease
* Inability (cognitively) to comprehend the instructions given during the trial and to comply with them

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Horizontal Intermediate Visual Field | Baseline
Visual Acuity | Baseline
Horizontal Near Visual Field | Baseline
Field of comfortable reading on a computer screen | Baseline
Horizontal Far Visual Field | Baseline

SECONDARY OUTCOMES:
Subjective Evaluation of Visual Quality | 2-3 weeks
Overall Subjective Feedback | 2-3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yosef Pikel, M.D, Principal Investigator — Ziv Medical Center, Zefat, Israel